CLINICAL TRIAL: NCT01503034
Title: Study of Tumor Characteristics, Patient Care and Prognosis of Women With Breast Cancer During a Pregnancy Diagnosed Between 2000 and 2014
Brief Title: Pregnant Women With a Breast Cancer Diagnosed Between 2000 and 2014
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: Cancer et grossesse
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Pregnant women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study cohort: This cohort is made up of pregnant women with a breast cancer diagnosed between 2000 and 2014.
- Compared cohort: This cohort is made up of non-pregnant women with a breast cancer diagnosed between 2000 and 2009.

SUMMARY:
This is a non-interventional, retrospective, multicentre study involving women having had a breast cancer during their pregnancy, diagnosed between 2000 and 2014 (cases) and non-pregnant women having had a breast cancer between 2000 and 2009 (controls).

DETAILED DESCRIPTION:
Investigators will explain the purpose of the study to the eligible patients, still alive, and will inform them verbally and in writing, using the information note, of their possibility of refusal. No information will be made for deceased patients.

The investigators will complete the case report forms on paper and then will send them by mail.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over
* Confirmed histological diagnosis of invasive breast cancer
* No known metastasis
* For the cases :

  * Patients pregnant at the time of the first diagnosis
  * 1st diagnosis between 2000 and 2014
* For the controls :

  * Patients not pregnant at the time of the first diagnosis
  * 1st diagnosis between 2000 and 2009

Exclusion Criteria:

* Patients who have undergone an induced abortion after the diagnosis of breast cancer
* Patients with a history of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study being retrospective, we will include all the subjects that meet our inclusion criteria over the period analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2010-12-14 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The overall survival corresponds to the time elapsed between the breast cancer diagnostic date and the death date.

SECONDARY OUTCOMES:
the support of breast cancer cases occured during pregnancy | 5 years
  Description of the anti-tumor treatment (surgery, radiotherapy, chemotherapy, hormone therapy, targeted therapy), of the imaging performed and of the childbirth (programmed or not, vaginal or caesarean section, baby's condition at birth, etc.).
Tumor characteristics | 5 years
  Description of the tumor characteristics on the diagnostic biopsy or on the surgical specimen : histological type, Her2 status, hormone receptor status, etc.
Disease-free survival | 5 years
  The disease-free survival is calculated from the time elapsed between the breast cancer diagnostic date and the first recurrence of the disease.
Case-control comparison | 5 years
  Comparison of the tumoral characteristics, the patient care and the prognosis of women with breast cancer appeared during a pregnancy, with non-pregnant women of the same age.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence VANLEMMENS, MD, Principal Investigator — Centre Oscar Lambret
Locations (37):
- France (37):
  - Clinique Sainte Catherine, Avignon
  - Cabinet Dr Le Guen Naas, Baud
  - Centre Hospitalier Universitaire, Besançon
  - Institut Bergonié, Bordeaux
  - CHR, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léonard de Vinci, Dechy
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre de Pharmacovigilance, Lille
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHRU La Peyronie et Centre Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Polyclinique de Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Radiologique, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Régaud, Toulouse
  - Cabinet Dr Leroy, Tourcoing
  - Hôpital Bretonneau - Centre régional de cancérologie Henry Kaplan, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif